CLINICAL TRIAL: NCT05367804
Title: Växtbaserade Proteiner påverkan på människors tarmhälsa Dietary Protein Impact on Human Gut Health
Brief Title: Dietary Protein Impact on Human Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PanProtein
Record Dates: First submitted 2022-03-17; First posted 2022-05-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Healthy male and female adult subjects (n=39) will be recruited to take part in an evaluation study to determine the amount of dietary protein intake which influences gut-protein-derived metabolites production. The study consists of 8 weeks with weekly visits and the subjects will consume an isolated plant-protein for 4 weeks (week 4 to 8), in each week the amount of protein supplementation will increase. Faecal samples will be used to answer the main outcome of gut metabolites and microbiota profile. And the blood and urine samples to measure health status and compliance (protein intake markers). Questionnaires will be used to access gastrointestinal symptoms and bowel movement, physical activity level and dietary intake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isolated plant protein (Experimental): Visit 1 to 8 participants will collect faecal samples. Visits 4 to 8 in addition to the faecal sample, urinary samples (24 h urine collection) will be collected by themselves, and blood sample will be collected at the hospital. For the visits with blood collection (visits 4 to 8), subjects will come to the study centre after 10 hours of overnight fast. Subjects will have anthropometry measurements taken in the visits 4, 5, 6, and 7 using a Tanita® full body composition. Subjects will respond to questionnaires about their physical activity (once a week), Gastrointestinal Symptom rating scale (GSRS - once a week) and track their intestinal habits using Bristol scale (every day). Subjects' diet will be assessed using a web-based 24-hour diet recall (interviewed so the participants learn how to use the tool regardless of where they are) followed by multiple day records (3 times a week).
  Interventions: Dietary Supplement: Isolated pea protein

INTERVENTIONS:
Dietary Supplement: Isolated pea protein — The subjects eligible to take part in this study will consume an isolated plant protein for 4 weeks (week 4 to 8), in each week the amount of protein supplementation will increase (0.25 to 1.0 g of protein per kg of body weight). The protein will be provided as a powder in opaque bags and participants will be instructed to dissolve the contained powder in liquids (as water) or on their food (e.g., yogurt, oat porridge). The baseline will consist of 4 visits (1 to 4) to see how stable are the baseline results.

SUMMARY:
The overall aim of this project is to evaluate the quantity of dietary protein that affects gut protein metabolization and if the baseline measurements are stable.

DETAILED DESCRIPTION:
Healthy male and female adult subjects (n=39) will be recruited to take part in an evaluation study to determine the amount of dietary protein intake which influences gut-protein-derived metabolites production. The subjects eligible to take part in this study will consume an isolated plant protein for 4 weeks, in each week the amount of protein supplementation will increase. The protein will be provided as a powder in opaque bags and participants will be instructed to dissolve the contained powder in liquids (as water) or on their food (e.g., yogurt, oat porridge). The baseline will consist in 4 visits, which in all visits faecal samples will be collected by themselves at their house or at hospital, using materials provided by the study staff. In one baseline visits (visit 4) in addition to the faecal sample, urinary sample will be collected by themselves, and blood samples will be collected at the hospital. After that, subjects will have the dietary intervention for four weeks and more 4 visits. For the visits with blood collection (visits 4 to 8), subjects will come to the study centre after 10 hours overnight fast. Subjects will have anthropometry measurements taken in the visits 4, 5, 6, and 7 using a Tanita® full body composition. Subjects will respond to questionnaires about their physical activity (once a week), Gastrointestinal Symptom rating scale (GSRS - once a week) and track their intestinal habits using Bristol scale (every day). Subjects' diet will be assessed using a web-based 24-hour diet recall (interviewed so the participants learn how to use the tool regardless of where they are) followed by multiple day records (3 times week).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Body mass index (BMI) 18,5-30 kg/m2
* Weight stable within the previous 3 months
* Maintenance of the usual physical activity habits during the study
* Intake of fibre between 15 and 25 g per day (evaluated by 3 food diaries or 24-hours recalls)
* Omnivores

Exclusion Criteria:

* Acute chronic disease, inflammatory or functional gastrointestinal diseases and any other disease or disorder that could affect the outcome of the study
* Use of a medication that may interfere the study outcome
* Eating disorder
* High protein intake (more than 15% of energy or maximum 1,2 g of protein per kg of body weight per day; evaluated by 3 food diaries or 24-hours recalls)
* Use of antibiotic medication during the last 3 months prior the first visit
* Use of antibiotic medication very early in life (e.g., asthmatic children or ear inflammation)
* Use of laxative or anti-diarrhoea medication within the past 3 months before the study
* Regular consumption of probiotic or prebiotic product for the past 6 weeks before the study
* Special diet that is considered to affect the study participation and/or study results, for example, high protein diets
* More than 5 h of moderate-vigorous exercise per week
* Pregnancy or breastfeeding
* Intolerance to dietary supplements that will be used in the study
* Smoking
* Abuse of alcohol or drugs (according to AUDIT score)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in the faecal metabolites using targeted and untargeted metabolomics | 8 weeks
  Difference in faecal metabolites depending on the protein supplementation amount. Targeted and untargeted metabolomics measurements will be used (e.g., short-chain fatty acids and branched chain fatty acids analyses, and polar and non polar metabolomics). Faecal samples will have their metabolites extracted and quantified by liquid chromatography coupled with high-resolution time-of-flight mass spectrometry (UHPLC-qToF-MS), and gas chromatography coupled with high-resolution mass spectroscopy (GC-Orbitrap). The level of metabolites will be compared throughout the whole study.
Routinely analysed markers for protein intake/compliance - urine | 5 weeks
  Difference in 24 h urine samples markers due to the protein supplementation (e.g., for 24 h urine: urea nitrogen from 24 h urine, creatinine, uric acid)
Routinely analysed markers for protein intake/compliance - blood | 5 weeks
  Difference in blood (serum) samples markers due to the protein supplementation (e.g., urea and creatinine)

SECONDARY OUTCOMES:
Food intake using food diaries | 8 weeks
  Food diaries 3 times a week
Changes in the gut microbiota profile during the baseline period | 4 weeks
  Difference in the gut microbiota profile/composition during the baseline period will be assessed by 16s/NGS (next-generation sequencing). Alpha and Beta diversity will be measured and compared throughout these 4 weeks of baseline.
Changes in the faecal metabolites during the baseline period | 4 weeks
  The difference in the metabolites profile during the baseline will be assessed by targeted and untargeted metabolomics. Targeted and untargeted metabolomics measurements will be used (e.g., short-chain fatty acids and branched chain fatty acids analyses and polar and non-polar metabolomics). Faecal samples will have their metabolites extracted and quantified by liquid chromatography coupled with high-resolution time-of-flight mass spectrometry (UHPLC-qToF-MS), and gas chromatography coupled with high-resolution mass spectroscopy (GC-Orbitrap). The level of metabolites will be compared during the baseline period.
Profile/composition of the gut microbiota during the intervention | 5 weeks
  Difference in the gut microbiota profile/composition because of the protein supplementation will be assessed by 16s/NGS. Alpha and Beta diversity will be measured and compared throughout the 5 weeks of intervention.
Assessment of the Gastrointestinal Symptom rating scale (GSRS) during the study | 8 weeks
  The gastrointestinal symptoms will be assessed during the baseline and protein supplementation period. Difference in the frequency and severity of gastrointestinal symptoms during the study will be assessed (15 questions with a scale of 1-7, minimum value 1, maximum 7, higher score correspond to a worse outcome)
Assessment of the bowel movement using the Bristol scale diary | 8 weeks
  The bowel movement will be assessed during the baseline and protein supplementation period by the Bristol scale diary. In the diary they write down the type of stool based on the scale which shows 7 pictures of different forms of stool, from watery diarrhea to compact. Participants are asked to choose the form of stool they have every day during the study.
Assessment of physical activity level | 8 weeks
  To assess the maintenance or difference of physical activity level during the baseline and dietary intervention by the AKTIVITETSVANOR questionnaire (Swedish questionnaire to assess physical activity frequency for 7 days).
Assessment of height | 5 weeks
  The height will be assessed in meters.
Assessment of body composition | 6 weeks
  Participants will be have their body composition measured using Tanita® full body scale. For this their height (m) will be measured and the information will be entered at the Tanita® scale. The obtained results by Tanita are: weight (kg), muscle mass (% and kg), body water content (% and kg), fat mass (% and kg), basal energy expenditure (kcal and kJ) and BMI in kg/m^2.
Assessment of body weight during the study | 6 weeks
  Participants will be weighted in order to have information of their body weight changes in kilograms during the study.
Concentrations of faecal calprotectin | 5 weeks
  Difference in faecal levels of calprotectin during the study intervention
Concentration of glucose | 5 weeks
  Measurement of glucose in blood samples
Concentration of insulin | 5 weeks
  Measurement of insulin in blood samples
Concentration of C-reactive protein | 5 weeks
  Measurement of C-reactive protein in blood samples
Concentration of cholesterol (total, LDL, and HDL) | 5 weeks
  Measurement of cholesterol (total, LDL, and HDL) in blood samples
Concentration of triglycerides | 5 weeks
  Measurement of triglycerides in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jan Brummer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Campus USÖ, Örebro University, Örebro, Sweden